CLINICAL TRIAL: NCT03900390
Title: The Study of Potency of Cross-preconditioning to Prevent Ischemic-reperfusion Injury for Heart Transplantation Recipient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mengya Liang (Other)
Responsible Party: Sponsor-Investigator, Mengya Liang, associate professor, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FirstSunYetSen118
Record Dates: First submitted 2019-03-04; First posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-03

CONDITIONS: Ischemic Preconditioning
Keywords: heart transplantation; ischemia-reperfusion injury
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cross Ischemic Preconditioning Group (Experimental): the ascending aorta of the CIP group will be crossclamped to cease the blood supply for 2 minutes, separated by a 3-minute rest interval, and repeated successively on 2 occasions
  Interventions: Procedure: cross-preconditioning
- Control Group (No Intervention): The recipients in the control group are to undergo routine cardiopulmonary bypass procedure of heart transplantation without Ischemic Preconditioning manoeuvre.

INTERVENTIONS:
Procedure: cross-preconditioning — After the establishment of the cardiopulmonary bypass, the ascending aorta of the CICP group will be crossclamped 2 minutes, separated by a 3-minute rest interval, and repeated successively on 2 occasions.
  Arms: Cross Ischemic Preconditioning Group

SUMMARY:
In recent years, a large number of studies confirmed the protective effect of ischemic preconditioning on myocardium against ischemia/reperfusion injury, but the clinical data of the effectiveness of ischemic preconditioning in heart transplantation is still missing. Inspired by the promising data of ischemic preconditioning from the previous reports, the investigators firstly introduce a novel method of cross ischemic preconditioning technique to prevent ischemia/reperfusion injury to heart transplant recipients.

This study will evaluate whether this cross-preconditioning technique would attenuate ischemia/ reperfusion injury to the heart transplant recipients, reduce Intensive Care Unit(ICU) and total hospitalization stays and the incidence of cardiovascular adverse events and improve the long-term survival outcomes.

DETAILED DESCRIPTION:
Patients receiving heart transplantation are randomly assigned into the cross ischemic preconditioning (CICP) intervention group and the control group. (the Statistical Analysis System (SAS) software was used to generate a random number table and randomly divided into two groups). After the establishment of the cardiopulmonary bypass, the ascending aorta of the CICP group will be crossclamped 2 minutes, separated by a 3-minute rest interval, and repeated successively on 2 occasions.

The recipients in the control group are to undergo routine cardiopulmonary bypass procedure of heart transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent heart transplantation；
2. Signed informed consent.

Exclusion Criteria:

1. Systemic active infection;
2. Refractory respiratory failure or renal failure;
3. Severe systemic diseases with limited survival time.
4. ABO blood groups incompatibility
5. positive serum HIV antibody;
6. drug or alcohol abusing;
7. Mentally ill;
8. Recent history of severe pulmonary embolism
9. Have not signed informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-07-07 (Actual); Primary Completion 2022-07-07 (Estimated); Study Completion 2023-07-07 (Estimated)

PRIMARY OUTCOMES:
serum troponin T/ creatine kinase-MB level | 3days
  troponin T/ creatine kinase-MB at definitive time points ( baseline, crossclamping, reperfusion, 6,24,48 and 72 hours postoperatively)
Number of Participants with major adverse cardiacand cerebrovascular events (MACCE) in one year postoperatively | 1year
  MACCE include death from cardiovascular causes, nonfatal myocardial infarction, coronary revascularization, or strok

SECONDARY OUTCOMES:
inotrope score | 3days
  calculated from the maximum dose of the individual inotropic agents administered in the first 3 days after surgery
serum creatinine level | 3days
  grade 1, 2, or 3 acute kidney injury within 72 hours after surgery (assessed on the basis of the increase in the serum creatinine level according to the International Kidney Disease: Improving Global Outcomes classification
ICU time | up to 2 weeks
  duration of stay in the intensive care unit and hospital
6-minute walk test | 2weeks
  distance on the 6-minute walk test two weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Zhongkai Wu, Study Director — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The first affiliated hospital of sun yat-sen university, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No